CLINICAL TRIAL: NCT01299584
Title: A Post Marketing Surveillance to Monitor the Safety of ULTIVA (Remifentanil) Adminstered in Korean Subjects According to the Prescribing Information
Brief Title: ULTIVA Post Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 105936
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Remifentanil: Patients administrated remifentanil at the site
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Basically there is no treatment allocation. Subjects who would be administered of remifentanil at their physicians' discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
This study is a post-marketing surveillance to monitor safety and efficacy of remifentanil during various surgeries and identify SAEs, adverse drug reactions, and unexpected AEs not described as precautions or warnings and to identify prognostic factors that have an effect on the AEs and to assess effectiveness of remifentanil in real clinical practices after marketing.

The subjects are patients prescribed for remifentanil by the investigators at the sites based on prescription information in normal clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anesthesia

Exclusion Criteria:

* According to precautions or warnings on PI, remifentanil should not be administered to the following patients
* Patients with any allergic reaction to any ingredients of remifentanil or other fentanyl analogues

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects are patients prescribed for Remifentanil by the investigators at the sites based on prescription information in normal clinical practices.
Sampling Method: Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2005-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this post-marketing surveillance (PMS) study was to monitor the safety and efficacy of Ultiva in the real clinical setting after launch.
Groups:
- Ultiva 1, 2, or 3 mg: One vial of Ultiva 1, 2, or 3 milligrams (mg) contains remifentanil hydrochloride (in-house specification) 1.10 mg, 2.21 mg, or 5.53 mg, respectively (as remifentanil 1 mg, 2 mg, or 5 mg, respectively). Participants were administered doses according to physician decision.
Period: Overall Study
Arm/Group | Ultiva 1, 2, or 3 mg
Started | 775
Completed | 766
Not Completed | 9
Not completed — Protocol Violation | 9

BASELINE CHARACTERISTICS:
Arm/Group | Ultiva 1, 2, or 3 mg
Number analyzed (Participants) | 766
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  Years | 45.3 (16.5)
Sex/Gender, Customized [Number; unit: Participants] — Baseline characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments. Gender data are missing for one participant.
  Participants
    Female | 422
    Male | 343
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  participants
    Korean | 766
    Not Korean | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Unexpected Serious Adverse Event
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. An unexpected event is an event that is not listed in the approval product information and is not described as a precaution or warning.
Time Frame: 24 hours
Population: Intent-to-Treat (ITT) Population: all participants who had been administered the investigational drug at least once and had undergone all safety assessments
Measure: Number; unit: participants
Arm/Group | Ultiva 1, 2, or 3 mg
Number analyzed (Participants) | 766
participants
  Participants with unexpected SAEs | 0
  Participants with no unexpected SAEs | 766

2. Secondary Outcome: Number of Participants With an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. For a list of all AEs occurring during the course of the study, see the table entitled "Other (Non-Serious) Adverse Events" in the Adverse Event section of the results record.
Time Frame: 24 hours
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Ultiva 1, 2, or 3 mg
Number analyzed (Participants) | 766
participants | 187

3. Secondary Outcome: Number of Participants With a Serious Adverse Event
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. For a list of all SAEs occurring during the course of the study, see the table entitled "Serious Adverse Events" in the Adverse Event section of the results record.
Time Frame: 24 hours
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Ultiva 1, 2, or 3 mg
Number analyzed (Participants) | 766
participants | 0

4. Secondary Outcome: Number of Participants With the Indicated Unexpected Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unexpected adverse events include those not listed in the approval product information and not described as precautions or warnings.
Time Frame: 24 hours
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Ultiva 1, 2, or 3 mg
Number analyzed (Participants) | 766
participants
  Dizziness | 1
  Chest discomfort | 1
  Dyspepsia | 1
  Headache | 1
  Dysuria | 1
  Coughing | 1
  Premature ventricular contraction | 1

ADVERSE EVENTS:
Description: Adverse events were coded by using World Health Organization Adverse Reactions Terminology (WHOART, preferred term level) according to the local regulation.
Arm/Group | Ultiva 1, 2, or 3 mg
Serious Adverse Events (participants affected / at risk) | 0/766
Other Adverse Events (participants affected / at risk) | 187/766
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultiva 1, 2, or 3 mg (N=766)
Hypotension (Cardiac disorders) | 123
Bradyarrhythmia (Cardiac disorders) | 105
Premature ventricular contraction (Cardiac disorders) | 1
Gagging (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Tremor after operation (General disorders) | 8
Chest discomfort (General disorders) | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 5
Coughing (Respiratory, thoracic and mediastinal disorders) | 1
Skeletal muscle stiffness (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Sedation (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.